CLINICAL TRIAL: NCT02762656
Title: The Effect of Perioperative Lidocaine Intravenous Infusion on Postoperative Recovery After Spine Surgery.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-16-2972-VS-CTIL
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Spinal Diseases
MeSH Terms: conditions — Spinal Diseases | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Patients will receive Lidocaine drip during spine surgery
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Patients will receive placebo during spine surgery
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine drip during surgery

SUMMARY:
The purpose of this study is to evaluate the effectiveness of perioperative Lidocaine intravenous infusion in reducing postoperative pain for spine surgery patients.

DETAILED DESCRIPTION:
Study design: this study used a prospective, randomized, double-blinded, and placebo-controlled clinical trial.

Sixty patients scheduled for a spine surgery will be randomly assigned to two groups. Lidocaine group will receive an intravenous bolus injection of lidocaine 1.5 mg/kg before intubation, followed by 2 mg/kg/h continuous infusion during the operation. Placebo group will receive the same dosage of saline at the same time. Analgesic requirement will be monitored using patient-controlled Analgesia (PCA protocol: demand dose is 2 mg of morphine, lockout 5 min, maximum dose 15 mg per hour). Forty-eight hours after surgery, we will check the morphine consumption in two groups. Quality of recovery after surgery will be assessed using Q0R15 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* spine surgery with general anesthesia

Exclusion Criteria:

* lidocaine allergy
* hepatic disease
* dementia or cognitive decline

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours postop
  Quality of recovery after surgery will be assessed using Q0R15 questionnaire and analgesic requirement will be monitored using PCA

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Intraoperative systemic infusion of lidocaine reduces postoperative pain after lumbar surgery: a double-blinded, randomized, placebo-controlled clinical trial. — http://www.ncbi.nlm.nih.gov/pubmed/24216403
- See also: Intravenous lidocaine for effective pain relief after a laparoscopic colectomy: a prospective, randomized, double-blind, placebo-controlled study. — http://www.ncbi.nlm.nih.gov/pubmed/25785316
- See also: Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. — http://www.cochrane.org/CD009642/ANAESTH_intravenous-infusion-lidocaine-starting-time-surgery-reduction-pain-and-improvement-recovery-after